CLINICAL TRIAL: NCT04267172
Title: A Prospective Randomised Controlled Study Assessing the Impact of Simulation Training in Primary Total Hip Replacement (THR).
Brief Title: Total Hip Replacement Performance & Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Buckinghamshire Healthcare NHS Trust (Other); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 270167
Record Dates: First submitted 2019-11-07; First posted 2020-02-12 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-01

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: The intervention to be tested is the simulation-based training and cognitive learning package. This will be delivered for 1-2 hours per week over a 4-week period in a supervised non-clinical setting to a randomised sub-group of 50% of the Surgical Residents enrolled into this study.
Who Masked: Outcomes Assessor
Masking Description: Consultant assessors will be blinded to the grouping of the Surgical Residents (additional simulation training group, or control group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Surgical Residents with additional simulation training (Experimental): Surgeon participant Group 1a: Interventional group ('StR's'): Trauma & Orthopaedic Specialty Registrars (Surgical Residents) on Arthroplasty clinical placements (n=6-8) receiving additional simulation training.
  Interventions: Behavioral: Surgical simulation training in primary Total Hip Arthroplasty
- Surgical Residents with routine training (Active Comparator): Surgeon participant Group 1b: control group (StR's): Trauma & Orthopaedic Specialty Registrars (Surgical Residents) on Arthroplasty clinical placements (n=6-8) receiving routine and normal training.
  Interventions: Other: No intervention: Surgical Resident Control Group
- Orthopaedic Surgeon 'Experts & Fellows' (Active Comparator): Consultant Orthopaedic Surgeons (n=5), and nationally appointed Arthroplasty Fellows (n=8). Surgeon participants within this group will not undergo any interventions.
  Interventions: Other: No Intervention: Consultant and Fellow Comparator Group

INTERVENTIONS:
Behavioral: Surgical simulation training in primary Total Hip Arthroplasty — The simulation-based and cognitive learning package will be delivered to a randomised sub-group of 50% of the Surgical Residents recruited into this study. This will be delivered in a supervised non-clinical setting within a dedicated University-owned simulation laboratory over a 4-week period for between 1 to 2 hours per week, over 3 to 4 consecutive but separate six-month placements.
  Arms: Surgical Residents with additional simulation training
Other: No intervention: Surgical Resident Control Group — Control Group
  Arms: Surgical Residents with routine training
Other: No Intervention: Consultant and Fellow Comparator Group — Comparator Group
  Arms: Orthopaedic Surgeon 'Experts & Fellows'

SUMMARY:
This research study is focused upon assessing and optimising surgeon's performance during, and patient outcomes following, primary total hip replacement (THR) surgery. The primary research question is to determine if additional simulation training can improve the intra-operative performance of surgical trainees (Residents) during a THR, or the outcome of patients after their THR. The investigators will aim to define an 'expert' standard in performing a primary elective THR, which may be used as a benchmark when assessing surgical trainee performance; and also determine if operative surgeon performance metrics during a THR are correlated with surgical experience, or patient outcomes.

DETAILED DESCRIPTION:
The surgeon participants in this study will be divided into 2 groups depending upon their position and seniority. The 'Expert' group will be composed of Consultant Orthopaedic Surgeons and Senior Fellows, and the 'Trainee' group will be composed of Trauma & Orthopaedic Specialty Registrars (Residents) on clinical placements in Adult Arthroplasty.

The intervention to be tested is the simulation-based training and cognitive learning package. This will be delivered for 1-2 hours per week over a 4-week period in a supervised non-clinical setting to a randomised sub-group of 50% of the Surgical Trainees enrolled into this study. Surgeon participants within the Expert/Fellow comparator group will not undergo any interventions.

The outcome measures will be surgeon-specific and patient-specific. These outcome measures for the 'Trainee' group will commence following completion of the simulation training (if applicable), whereas they can commence immediately following study approval for the 'Expert' group. The surgeon-specific outcome measures will be the objective motion-analysis metrics generated by validated and extensively used wireless sensors placed on the elbows of surgeons under their sterile gowns during the operation; and subjective assessments of surgical trainee performance using validated and reliable forms of structured human grading. Patient-specific outcome measures will be collected for a pre-determined number of patients who have undergone a primary elective THR by any of the surgeon participants in this study. All patient participants will be asked to provide their written informed consent for the use of their data in this study. The patient-specific outcome measures include: pre- and post-operative blood tests and radiograph (X-ray) analysis; the incidence of blood transfusions and any other peri-operative complications; the in-patient length of stay; and two patient-reported outcome measure (PROMs) questionnaires, namely the Oxford Hip Score (OHS) and EQ-5D.

Statistical analysis will be performed on the data collected, specifically aiming to identify any significant differences in either surgeon performance metrics, or patient outcome measures between:

1. The Surgical Trainees who have undertaken additional simulation training versus those who have routine training.
2. The 'Trainee' group and the 'Expert' group. A sub-group analysis may be performed within the 'Expert' group also to determine any differences between the Consultants and Fellows.

In summary, this novel research will use validated methodology and routinely collected patient outcome measures in order to determine the impact of simulation training on surgical trainee performance and patient outcomes following a primary elective THR, and also help to benchmark an expert level of performance in this commonly performed and highly effective operation. The results of this study will hopefully help in shaping the future of orthopaedic surgical training and assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with primary hip osteoarthritis who have been listed for elective primary Total Hip Replacement within the United Kingdoms National Health Service.
* Total Hip Replacement performed by a surgeon participant as lead surgeon.

Exclusion Criteria:

* Patients with complex hip pathology (e.g. previous trauma, hip dysplasia, infection).
* Patients who have had previous surgery on their affected hip.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Botnar Research Centre, Oxford, Oxfordshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number of patients recruited exceeded the number in protocol enrolment as it was necessary to continue patient recruitment within the Resident Groups to achieve the required number to power the primary outcome (i.e. operative time, n=25 in group 1a and 1b).
Groups:
- Surgical Residents With Additional Simulation Training: Surgeon participant Group 1a: Interventional group ('StR's'): Trauma & Orthopaedic Specialty Registrars (Surgical Residents) on Arthroplasty clinical placements (n=4) receiving additional simulation training.
  The intervention tested in this study was a one-day intensive simulation-based training module which was delivered to a randomised sub-group of surgeon participants within the 'novice' group.
- Surgical Residents With Routine Training: Surgeon participant Group 1b: control group (StR's): Trauma & Orthopaedic Specialty Registrars (Surgical Residents) on Arthroplasty clinical placements (n=3) receiving routine and normal training.
  No intervention: Surgical Resident Control Group: Control Group
- Orthopaedic Surgeon 'Experts & Fellows': Consultant Orthopaedic Surgeons (n=8), and nationally appointed Arthroplasty Fellows (n=8). Surgeon participants within this group will not undergo any interventions.
- Surgical Residents With Additional Simulation Training - Patients: Recruited Patients undergoing primary Total Hip Replacement by Surgical Residents With Additional Simulation Training.
- Surgical Residents With Routine Training - Patients: Recruited Patients undergoing primary Total Hip Replacement by Surgical Residents With Routine Surgical Training.
- Orthopaedic Surgeon 'Experts & Fellows' - Patients: Recruited Patients undergoing primary Total Hip Replacement by Arthroplasty Fellows or Consultants.
Period: Overall Study
Arm/Group | Surgical Residents With Additional Simulation Training | Surgical Residents With Routine Training | Orthopaedic Surgeon 'Experts & Fellows' | Surgical Residents With Additional Simulation Training - Patients | Surgical Residents With Routine Training - Patients | Orthopaedic Surgeon 'Experts & Fellows' - Patients
Started | 4 | 3 | 16 | 25 | 27 | 168
Completed | 4 | 3 | 16 | 25 | 27 | 168
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Surgical Residents With Additional Simulation Training - Patients",: Patients recruited into the study with operation led by surgical residents with additional simulation training (Group 1a)
- "Surgical Residents With Routine Training - Patients",: Patients recruited into the study with operation led by surgical residents without additional simulation training (Group 1b)
- "Orthopaedic Surgeon 'Experts & Fellows' - Patients": Patients recruited into the study with operation led by Arthroplasty Fellows or Consultants.
- Total: Total of all reporting groups
Arm/Group | Surgical Residents With Additional Simulation Training | Surgical Residents With Routine Training | Orthopaedic Surgeon 'Experts & Fellows' | Surgical Residents With Additional Simulation Training - Patients", | "Surgical Residents With Routine Training - Patients", | "Orthopaedic Surgeon 'Experts & Fellows' - Patients" | Total
Number analyzed (Participants) | 4 | 3 | 16 | 25 | 27 | 168 | 243
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 16 | 7 | 6 | 51 | 87
  >=65 years | 0 | 0 | 0 | 18 | 21 | 117 | 156
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 21 | 23 | 109 | 154
  Male | 3 | 3 | 16 | 4 | 4 | 59 | 89
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 16 | 0 | 0 | 0 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 25 | 27 | 168 | 220
Region of Enrollment [Number; unit: participants]
  United Kingdom | 4 | 3 | 16 | 25 | 27 | 168 | 243

OUTCOME MEASURES:

1. Primary Outcome: Surgeon Participant Intra-operative Motion Analysis
Description: Total number of surgeon hand movements obtained from elbow worn wireless motion sensors for each operation performed by the recruited surgeon participant as lead surgeon.
Time Frame: Intra-operatively (single patient participant)
Population: Outcome measure results represent the group mean average and standard deviations.
  Only Surgeon participants were assessed.
Measure: Mean (Standard Deviation); unit: Movement counts
Arm/Group | Surgical Residents With Additional Simulation Training | Surgical Residents With Routine Training | Orthopaedic Surgeon 'Experts & Fellows'
Number analyzed (Participants) | 4 | 3 | 16
Movement counts | 171,967 (41,867) | 172,258 (43,300) | 150,505 (38,190)

2. Primary Outcome: Surgeon Participant Intra-operative Timings
Description: Total time taken by each surgeon participant per step of the total hip replacement for each operation performed as lead surgeon.
Time Frame: Intra-operatively (single patient participant)
Population: Outcome measure results represent the group mean average and standard deviations for total operative time.
  Only Surgeon participants were assessed.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Surgical Residents With Additional Simulation Training | Surgical Residents With Routine Training | Orthopaedic Surgeon 'Experts & Fellows'
Number analyzed (Participants) | 4 | 3 | 16
Seconds | 4948 (1119) | 4428 (1122) | 3679 (828)

3. Primary Outcome: Surgical Trainee Global Rating Scale (GRS)
Description: A subjective human grading assessment of surgical performance rated on a scale of 7-35 with a higher score indicating a better surgical performance. GRS only performed for group 1a and 1b (i.e. Residents). Expert group did not have GRS collected.
Time Frame: Assessment performed post-operatively within 60 minutes following procedure for each patient participant.
Population: Outcome measure results represent the group median average and interquartile ranges.
  Only Surgical Resident participants were assessed.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Surgical Residents With Additional Simulation Training | Surgical Residents With Routine Training
Number analyzed (Participants) | 4 | 3
score on a scale | 30 [23 to 33] | 31 [25 to 34.25]

4. Primary Outcome: Percent of Participants With 4+ Objective Structured Assessment of Technical Skills (OSATS) Rating.
Description: A subjective human grading assessment of surgical performance. Rated on a 5 point scale, with a higher score indicating a more competently performed procedure. OSATS only performed for group 1a and 1b (i.e. Residents). Expert group did not have OSATS collected.
Time Frame: Assessment performed post-operatively within 60 minutes following procedure for each patient participant.
Population: The OSAT used was a standardised, validated OSAT used by the joint committee of surgical training (JCST) in the UK.
  Only Surgical Resident participants were assessed.
Measure: Number; unit: % of participants achieving level 4 OSAT
Arm/Group | Surgical Residents With Additional Simulation Training | Surgical Residents With Routine Training
Number analyzed (Participants) | 4 | 3
% of participants achieving level 4 OSAT | 55.5 | 37.5

5. Secondary Outcome: Post-operative Patient X-ray
Description: Post-operative X-ray analysis for component orientation for each patient recruited into this study whose operation was performed by a recruited surgeon participant as lead surgeon.
Time Frame: Assessment performed post-operatively within 8 weeks following procedure for each patient participant.
Population: radiographic inclination of acetabular cup. Outcome measure results represent the group mean average and standard deviation.
  Only patient participants were assessed.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Surgical Residents With Additional Simulation Training - Patients. | Surgical Residents With Routine Training - Patients. | Orthopaedic Surgeon 'Experts & Fellows' - Patients.
Number analyzed (Participants) | 25 | 27 | 168
degrees | 42.2 (6.7) | 43.0 (7.7) | 41.9 (7.8)

6. Secondary Outcome: Patient Blood Loss.
Description: Estimated on-table blood loss (OTBL) for each patient participant whose operation performed by the recruited surgeon participant as lead surgeon.
  This figure was calculated by subtracting the total volume of intra-operative irrigation fluid used from the total volume of fluid in the suction canister in addition to weighing the surgical swabs.
Time Frame: Assessment performed post-operatively within 60 minutes following procedure for each patient participant.
Population: Outcome measure results represent the group mean average and standard deviations.
  Only patient participants were assessed.
Measure: Mean (Standard Deviation); unit: millilitres
Arm/Group | Surgical Residents With Additional Simulation Training - Patients. | Surgical Residents With Routine Training - Patients. | Orthopaedic Surgeon 'Experts & Fellows' - Patients.
Number analyzed (Participants) | 25 | 27 | 168
millilitres | 339 (170) | 274 (150) | 316 (202)

7. Secondary Outcome: Number of Participants Requiring a Blood Transfusion.
Description: The number of units of packed red blood cells transfused for each patient participant (if applicable).
Time Frame: Assessment performed per single patient participant during in-patient stay up to 14 days following operation.
Population: Blood transfusions required. Only patient participants were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical Residents With Additional Simulation Training - Patients. | Surgical Residents With Routine Training - Patients. | Orthopaedic Surgeon 'Experts & Fellows' - Patients.
Number analyzed (Participants) | 25 | 27 | 168
Participants | 0 | 1 | 1

8. Secondary Outcome: Patient Hospital Length of Stay
Description: Length of stay (total days) for each patient recruited into this study.
Time Frame: From post-operation through to hospital discharge.
Population: Length of post-operative in-patient stay (days). Outcome measure results represent the group mean average and standard deviation.
  Only patient participants were assessed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Surgical Residents With Additional Simulation Training - Patients. | Surgical Residents With Routine Training - Patients. | Orthopaedic Surgeon 'Experts & Fellows' - Patients.
Number analyzed (Participants) | 25 | 27 | 168
days | 2.95 (2.2) | 3.37 (2.59) | 2.41 (2.11)

9. Secondary Outcome: Oxford Hip Score
Description: A joint-specific patient-reported outcome measure (PROM) to be assessed pre- and post-operatively. This is a 12 item questionnaire scored on a scale of 0-48, with a higher score representing better joint function. The change in score is presented and is defined as the value of the later time point (3-4 months post-operatively) minus the value at the earlier time point (pre-operatively).
Time Frame: Determined for each recruited patient pre-operatively and again at 3-4 months post-operatively
Population: Change in OHS. Outcome measure results represent the group mean average and standard deviation.
  Only patient participants were assessed.
Measure: Mean (Standard Deviation); unit: Score on a scale.
Arm/Group | Surgical Residents With Additional Simulation Training - Patients. | Surgical Residents With Routine Training - Patients. | Orthopaedic Surgeon 'Experts & Fellows' - Patients.
Number analyzed (Participants) | 25 | 27 | 168
Score on a scale. | 26 (10) | 24 (8) | 25 (8)

10. Secondary Outcome: EQ-5D
Description: A general patient-reported outcome measure (PROM) to be assessed pre- and post-operatively. The EQ-5D is comprised of 5 short questions each rated on a scale of 1-5 (25 points in total), with a higher score indicating a higher quality of life, and a visual analogue scale (EQ VAS) from 0-100, with a higher score indicating better health. The change in score is presented and is defined as the value of the later time point (3-4 months post-operatively) minus the value at the earlier time point (pre-operatively).
Time Frame: Determined for each recruited patient pre-operatively and again at 3-4 months post-operatively.
Population: Change in EQ-5D VAS. Outcome measure results represent the group mean average and standard deviation.
  Only patient participants were assessed.
Measure: Mean (Standard Deviation); unit: Score on a scale.
Arm/Group | Surgical Residents With Additional Simulation Training - Patients. | Surgical Residents With Routine Training - Patients. | Orthopaedic Surgeon 'Experts & Fellows' - Patients.
Number analyzed (Participants) | 25 | 27 | 168
Score on a scale. | 19 (14) | 19 (16) | 19 (14)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Surgical Residents With Additional Simulation Training | Surgical Residents With Routine Training | Orthopaedic Surgeon 'Experts & Fellows' | Surgical Residents With Additional Simulation Training - Patients. | Surgical Residents With Routine Training - Patients. | Orthopaedic Surgeon 'Experts & Fellows' - Patients.
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/16 | 0/25 | 0/27 | 0/168
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/16 | 0/25 | 0/27 | 0/168
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/16 | 0/25 | 0/27 | 0/168

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT04267172/Prot_SAP_000.pdf
  • Informed Consent Form: Patient Consent (2019-10-12): https://cdn.clinicaltrials.gov/large-docs/72/NCT04267172/ICF_001.pdf
  • Informed Consent Form: Surgeon Consent: Residents (2019-10-12): https://cdn.clinicaltrials.gov/large-docs/72/NCT04267172/ICF_002.pdf
  • Informed Consent Form: Surgeon Consent: Fellows and Consultants (2019-10-12): https://cdn.clinicaltrials.gov/large-docs/72/NCT04267172/ICF_003.pdf